CLINICAL TRIAL: NCT01575912
Title: Past Pain Experience and Perception of Experimental Pain
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Dominique Malauzat, MD, Centre Hospitalier Esquirol
Other Study IDs: 2012-A00047-36
Record Dates: First submitted 2012-03-13; First posted 2012-04-12 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Schizophrenia; Major Depression
Keywords: Schizophrenia; Major depression; Pain; Past pain experience
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- schizophrenia SC: subjects with a diagnosis of schizophrenia (SC) according to the DSM-IV-TR, submitted to experimental pain tests
  Interventions: Other: experimental pain tests
- major depression MD: subjects with a diagnosis of major depression (MD) according to the DSM-IV-TR, submitted to experimental pain tests
  Interventions: Other: experimental pain tests
- controls C: subjects without any diagnosis of psychiatric disorder (C) submitted to experimental pain tests
  Interventions: Other: experimental pain tests

INTERVENTIONS:
Other: experimental pain tests

SUMMARY:
Differences in pain perception between subjects with and without psychiatric illness may be influenced by the individual experience, and not primarily by the pathology, although the pathological frame may amplify it.The aim of this study is to establish if the characteristics of experimental pain feeling are influenced by the past pain experience, anxiety and emotion, independently from the diagnosis. The pain experience will be evaluated by an inventory of the potentially painful situations that one can come across through the life, to determine the following points : Number of painful events in the past, number of painful points during the last 6 months, number of painful events lasting more than 6 months, sum of pain intensities (graduated with Visual Analogic Scale VAS from 0 to 10), sum of gravity (evaluated from 0 to 5), the category of pain experience qualification (mostly affective, mostly sensorial, or both).

Schizophrenic, depressed and control participants will be recruited, and their pain experience throughout life will be put it in relation to experimental pain tests results (pressure application, ischemia induction), anxiety and emotion (Hospital Anxiety and Depression scale HAD), catastrophizing (Pain Catastrophizing Scale PCS), Heart Rate (HR) variation, Blood Pressure (BP) variation.

DETAILED DESCRIPTION:
The perception of moderated experimental pain (about 3 out of ten with visual analogue scale VAS) in subjects with schizophrenia (Girard et coll., 2011), major depression (ED) (bipolar or isolated/recurrent episode) (to be published) in comparison with controls without psychiatric pathologies show that exploration of pain in situation like medical examination to identify painful points should be done in the same conditions for persons with psychiatric troubles and persons without mental disease. But the risk is that the expression of pain, either in experimental conditions nor in the daily life, is not in relation with the feeling or perception of pain. Numerous factors may interfere in the pain message modulation, like the past pain experience, stress and anxiety, which are not or partially explored in experimental studies. The individual experience of pain is constructed throughout the whole life, from several influences (biological, psychological, and sociocultural). The symptoms interfaces of the different psychiatric troubles seem to be widely involved in the pain process, and its progressive construction. This study aims to better understand the relationships between all those variables.

Procedures applied :

Anterior pain experience evaluation (questionnaire); Pain tests : 160 kPa pressure application to determine corresponding pain with VAS), and ischemia induction to determine the time necessary to obtain a pain equivalent to 3 out of 10; anxiety and emotional evaluation (Hospital Anxiety and Depression scale), catastrophizing evaluation (Pain Catastrophizing Scale), HR variation and BP variation (vegetative measures linked to anxiety) collection of diagnosis, and therapeutic treatment

ELIGIBILITY:
Inclusion Criteria:

* subjects with psychiatric trouble : diagnosis of schizophrenia or major depression according to the DSM-IV-TR criteria.
* control subjects : without known psychiatric history.
* age between 18 and 60.

Exclusion Criteria:

* absence of consent, hospitalization under constraint, absence of health insurance.
* inability to answer the questionnaires
* pregnancy
* antalgic or analgesic treatment
* allergy to latex
* non stabilized high blood pressure, bad blood coagulation,
* peripheral neuropathy, nerve lesion, dermatosis at the superior extremities, muscular lesion or pathology at the upper member level
* non treated alcohol dependence
* illegal substance consumption in the past 48 hours
* participation to an other biomedical study during the 2 weeks before inclusion, and until the pain tests, if this study can interfere with the realization of the objectives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects hospitalized in the Esquirol Hospital center with schizophrenia or major depression according to the DSM-IV-TR criteria.
  Subjects without without known psychiatric history. Recruited persons will be matched according to age classes.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Malauzat, MD, Principal Investigator — Centre Hospitalier Esquirol
Locations (1):
- Centre Hospitalier Esquirol, Limoges, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Girard M, Plansont B, Bonnabau H, Malauzat D. Experimental pain hypersensitivity in schizophrenic patients. Clin J Pain. 2011 Nov-Dec;27(9):790-5. doi: 10.1097/AJP.0b013e31821d904c. PMID 21593663

RESULTS

PARTICIPANT FLOW:
Groups:
- Group of Subjects Presenting Schizophrenia SC: subjects presenting a schizophrenia according to the DSM-IV-TR and submitted to experimental pain tests
- Group of Subjects Presenting Major Depression MD: subjects presenting a major depression according to the DSM-IV-TR and submitted to experimental pain tests
- Group of Subjects Without Psychiatric Troubles C: subjects without any psychiatric disorder and submitted to experimental pain tests
Period: Overall Study
Arm/Group | Group of Subjects Presenting Schizophrenia SC | Group of Subjects Presenting Major Depression MD | Group of Subjects Without Psychiatric Troubles C
Started | 30 | 32 | 30
Completed | 30 | 32 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group of Subjects With Schizophrenia SC: subjects presenting a schizophrenia according to the DSM-IV-TR and submitted to experimental pain tests
- Group of Controls Without Psychiatric Disorder: subjects without any psychiatric disorder and submitted to experimental pain tests
- Total: Total of all reporting groups
Arm/Group | Group of Subjects With Schizophrenia SC | Group of Subjects Presenting Major Depression MD | Group of Controls Without Psychiatric Disorder | Total
Number analyzed (Participants) | 30 | 32 | 30 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (9.72) | 44.69 (10.08) | 41.53 (10.27) | 43.21 (10.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 27 | 17 | 51
  Male | 23 | 5 | 13 | 41
Region of Enrollment [Number; unit: participants]
  France | 30 | 32 | 30 | 92

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale Evaluation for the Pre-fixed Pressure Test
Description: pain tests will be realized during the first week of hospitalization for the persons hospitalized for major depression, and during the period of hospitalization (after stabilization) for the persons presenting schizophrenia.
  The controls are tested within one month of the study information. total range : 0 - 10. The intensity of pain increases with the value of VAS. 10 corresponds to an unbearable pain.
Time Frame: one month
Population: analysis per arm group
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group of Subjects With Major Depression MD: subjects presenting a major depression according to the DSM-IV-TR and submitted to experimental pain tests
- Group of Subjects Without Psychiatric Troubles C: control subjects without any psychiatric disorder
Arm/Group | Group of Subjects Presenting Schizophrenia SC | Group of Subjects With Major Depression MD | Group of Subjects Without Psychiatric Troubles C
Number analyzed (Participants) | 30 | 32 | 30
units on a scale | 2.8 (3.2) | 2.1 (1.8) | 1.2 (1.3)
Statistical Analysis 1: Comparison: Group of Subjects Presenting Schizophrenia SC vs Group of Subjects With Major Depression MD vs Group of Subjects Without Psychiatric Troubles C; Test type: Other; p = 0.121, Wilcoxon (Mann-Whitney) — using Mann Whitney test

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Group of Subjects With Schizophrenia SC: subjects presenting a diagnosis of schizophrenia according to the DSM IV TR and submitted to experimental pain tests
- Group of Subjects Presenting Major Depression MD: subjects presenting a diagnosis of major depression according to the DSM IV TR and submitted to experimental pain tests
- Group of Controls Without Psychiatric Disorder: control subjects without any psychiatric disorder and submitted to experimental pain tests
Arm/Group | Group of Subjects With Schizophrenia SC | Group of Subjects Presenting Major Depression MD | Group of Controls Without Psychiatric Disorder
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/32 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes